CLINICAL TRIAL: NCT06592313
Title: Difficult Airway in the Bariatric Patient: The BARINTUBE Cohort Study
Acronym: BARINTUBE
Status: Completed | Type: Observational
Sponsor: : Manuel Alberto Guerrero Gutierrez (Other Government)
Responsible Party: Sponsor-Investigator, : Manuel Alberto Guerrero Gutierrez, Principal Investigator, Instituto Mexicano del Seguro Social
Organization: Instituto Mexicano del Seguro Social (Other Government)
Other Study IDs: 1667/17-05-2024
Record Dates: First submitted 2024-09-09; First posted 2024-09-19 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2026-01

CONDITIONS: Obesity; Bariatric Surgery Candidate
Keywords: bariatric surgery; difficult airway; videolaringoscopy; intubation; airway managment; obesity and anesthesia; preoperative care
MeSH Terms: conditions — Obesity | interventions — Intubation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients undergoing bariatric surgery: Adults with an indication for bariatric surgery who have been schedule for a bariatric surgery procedure.
  Interventions: Procedure: Intubation

INTERVENTIONS:
Procedure: Intubation — Aiway management procedure involving the Insertion of an orotracheal cannula through the oropharynx.

SUMMARY:
Background: Difficult airway in bariatric patients presents significant challenges during anesthesia, impacting patient safety and surgical outcomes. This study aims to estimate the incidence of difficult airway in bariatric patients undergoing surgery.

Materials and Methods: This prospective observational cohort study will be conducted in a single center. Patients over 18 years with a BMI ≥ 30 kg/m2 undergoing bariatric surgery and requiring intubation will be included. Data will be collected on patient demographics, clinical characteristics, and intubation outcomes. The primary outcome is the occurrence of difficult airway, defined by specific criteria including intubation difficulty and the need for alternative airway management techniques. Secondary outcomes include complications related to airway management and overall surgical outcomes. A total of 1290 patients will be included in the study to estimate the incidence of difficult airway within a confidence of 3%.

Conclusions: Difficult airway management in bariatric patients is relatively common and is influenced by specific patient factors. The findings of this study will mainly allow the estimation of difficult airway incidence in patients with bariatric surgery under the new clinical definitions.

ELIGIBILITY:
Inclusion Criteria:

* Patients over 18 years of age
* Patients of both genders
* Patients diagnosed with BMI greater than or equal to 30 kg/m2
* Patients who will undergo bariatric surgery
* Patients who require intubation for intraoperative ariway management

Exclusion Criteria:

* Patients who withdraw their consent to participate in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with a body mass index greater than or equal to 30 kg/m2 scheduled for bariatric surgery.
Sampling Method: Non-Probability Sample
Enrollment: 1290 (Actual)
Dates: Start 2024-10-15 (Actual); Primary Completion 2025-12-16 (Actual); Study Completion 2025-12-20 (Actual)

PRIMARY OUTCOMES:
Incidence of difficult airway | Day 1
  Cumulative incidence (expressed as a percentage), according to the American Society of Anesthesiologists 2022 definition of difficult airway (anticipated or unanticipated difficulty or failure is experienced by a physician trained in anesthesia care, including but not limited to one or more of the following: facemask ventilation, laryngoscopy, ventilation using a supraglottic airway, tracheal intubation, extubation, or invasive airway).

SECONDARY OUTCOMES:
Incidence of severe hypoxia | Day 1
  Cumulative incidence (expressed as percentage) of severe hypoxia, defined as a peripheral blood oxygen saturation (SpO2) lower than 80% during advanced airway management.
Incidence of cardiovascular collapse | Day 1
  Cumulative incidence (expressed as percentage) of cardiovascular collapse, defined as any of the following events within 30 minutes from induction to surgical incision:
  * Systolic blood pressure lower than 65 mmHg.
  * Dyastolic blood pressure ower than 90 mmHg for more than 15 minutes
  * Unplanned need for vasopressors or fluid loading greater than; 15 ml/kg to maintain target blood pressure.
Incidence of minor adverse events | Day 1
  Cumulative incidence (expressed as percentage) of minor adverse events, including:
  * Moderate hypoxia (SpO2 lower than 93%),
  * Airway injury,
  * Clinically relevant bleeding,
  * Oral aspiration of gastric contents,
  * Dental injury,
  * Lip injury.
Incidence of Difficult Facemask Ventilation | Day 1
  Cumulative incidence (expressed as a percentage), according to the American Society of Anesthesiologists 2022 definition of Difficult Facemask Ventilation (It is not possible to provide adequate ventilation, because of one or more of the following problems: inadequate mask seal, excessive gas leak, or excessive resistance to the ingress or egress of gas.). For operationalization, successful face mask ventilation with 2 hands will be consigned as the reference (No difficult face mask ventilation), whereas face mask ventilation attempts with 4 or 6 hands will be considered as the presence of difficult face mask ventilation.
Incidence of Difficult or Failed Tracheal Intubation | Day 1
  Cumulative incidence (expressed as a percentage), according to the American Society of Anesthesiologists 2022 definition of Difficult or Failed Tracheal Intubation (Tracheal intubation requires multiple attempts or tracheal intubation fails after multiple attempts.). For operationalization, more than 1 attempt will be considered as Difficult or Failed Tracheal Intubation.

OTHER OUTCOMES:
Predictors of Difficult Airway | Day 1
  Predictors of difficult airway will be identified through a multivariable generalized linear regression model.
Predictors of Difficult or Failed Tracheal Intubation | Day 1
  Predictors of greater number of intubation attempts will be identified through a multivariable generalized linear regression model.
Successful intubation rate according to laryngoscopy method | Day 1
  Participants will be grouped according to the laryngoscopy method (direct laryngoscopy vs videolaryngoscopy) and the cumulative incidence of successful intubation (expressed as proportion) will be calculated for each group. The risk difference and an appropriate measure of association (i.e., risk ratio, odds ratio) will be estimated.

CONTACTS AND LOCATIONS:
Locations (1):
- Centro Medico Bariatrico, Tijuana, Estado de Baja California, Mexico

IPD SHARING:
Plan to Share IPD: Yes
Anonymized individual participant data will be deposited and made available through an open acess data repository (i.e., Harvard Dataverse). Any potentially sensitive patient-identifying data will either not be released or will undergo minimization and aggregation/abstraction procedures to reduce participant identification risk. Informed consent forms will indicate that a minimal risk of re-identification cannot be excluded despite all these participant data protection methods,in compliance with current IPD sharing recommendations.
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Time Frame: IPD and supporting information will be made available with the final original research article, which will be made available as a preprint within a maximum 1-year term after the study conclusion date. This report will be subsequently sent for publication in a peer-reviewed journal. Other pre-specified outcomes may be reported in separate publication after the main research article, reason why the indicated time frame does not apply for such outcomes. There is not an anticipated end term for access to the data and supporting information, as these will be deposited in data and code repository sites as priorly indicated.
Access Criteria: No data and supporting information access restrictions are anticipated, as these will be deposited in open access repositories (i.e., Harvard Dataverse, Open Science Framework, Zenodo).